CLINICAL TRIAL: NCT01715558
Title: Clinical Outcome of Pacemaker paTIents According to Pacing Modality and Primary INDications
Brief Title: Clinical Outcome of Pacemaker paTIents According to Pacing Modality and Primary INDications OPTI-MIND 2
Acronym: OPTI-MIND 2
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM00053871 / 90942887
Record Dates: First submitted 2012-10-15; First posted 2012-10-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-02

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RYTHMIQ study group
- Historical control from OPTI-MIND

SUMMARY:
The purpose of the study is to demonstrate that reduction of unnecessary pacing provided by RYTHMIQ algorithm programed to ON in a pacemaker is associated with better clinical outcomes in bradycardia target population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients implanted with any of BSC dual chamber PM devices equipped with RHYTMIQ with the algorithm programed to ON based on clinical indication at the time of discharge from the hospital
2. Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center
3. Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Patients with 3rd degree AV block
2. Patients with permanent AF
3. Patients followed up remotely with remote patient management system.
4. Patients who are unable to be followed up by the participating centers for a period of two years
5. Patients who have a current device implanted for more than 15 days
6. Women of childbearing potential who are pregnant, or plan to become pregnant during the time of the study (method of assessment upon physician's discretion)
7. Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry or extensions/amendments of the current protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with permanent pacemaker with RYTHMIQ programed to ON
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Combined event rate of all-cause mortality, cardiovascular hospitalizations and atrial fibrillation at 2 years in a specific Brady population implanted with BSC PM devices equipped with RYHTMIQ feature | 2 years
  Combined event rate of all-cause mortality, cardiovascular hospitalizations and atrial fibrillation at 2 years in a specific Brady population implanted with BSC PM devices equipped with RYHTMIQ feature compared to data from a cohort of subjects implanted with BSC PM without RYTHMIQ pooled from OPTI-MIND study.

SECONDARY OUTCOMES:
Combined event rate of all-cause mortality, cardiovascular hospitalizations and atrial fibrillation at 2 years stratified per patient characteristics. | 2 years
  A multivariate model will be used to find the independent association with the combined primary endpoint, RYTHMIQ algorithm and other patient characteristics.
  Variables of interests include (but are not limited to): primary pacing indication (SND vs AVB), degree of AVB, age, gender, underlying disease, use of Betablockers, history of atrial fibrillation, LVEF, NYHA class, RV lead position, type of sensors used.

CONTACTS AND LOCATIONS:
Locations (39):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Hartcentrum Hasselt Jessa Ziekenhuis Campus Virga Jesse, Hasselt
- Denmark (3):
  - Regionshospitalet Herning, Herning
  - Vejle Sygehus, Vejle
  - Viborg Sygehus, Viborg
- France (8):
  - CHRU Angers, Angers
  - CHRU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble - Hopital Michallon, Grenoble
  - Hôpital la Roche sur Yon, La Roche-sur-Yon
  - Service de cardiologie, CHU Nancy-Brabois, Nancy
  - CHU de Nantes-Hopital Laennec, Nantes
  - Centre Hospitalier Général de Pau, Pau
  - CHU Poitiers - Hôpital La Miletrie, Poitiers
- Germany (4):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Universitätsklinikum, Leipzig
  - St.-Marien-Hospital GmbH, Lünen
  - Deutsches Herzzentrum München, München
- Italy (11):
  - Ospedale Cardinal Massaia, Asti
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Policlinico S. Orsola - Malpighi, Bologna
  - Pres. Osp. F. Ferrari, Casarano (LE)
  - Ospedale Civile San Leonardo, Castellammare di Stabia
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Ospedale Santa Maria degli Angeli, Pordenone
  - P.O. Santa Maria Delle Grazie, Pozzuoli
  - Ospedale "Misericordia e Dolce" - AZIENDA USL 4 PRATO, Prato
  - Azienda ospedaliera Sant'Andrea, Rome
  - Policlinico Tor Vergata, Rome
- Netherlands (4):
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Elisabeth Ziekenhuis, Tilburg
  - Gelre Ziekenhuis Zutphen, Zutphen
- Slovakia (2):
  - SUSCCH a.s., Banská Bystrica
  - The National Institute of Cardiovascular Diseases, Bratislava
- Spain (3):
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital San Pedro, Logroño
  - Hospital de Torrejón, Torrejón
- United Kingdom (2):
  - Blackpool Victoria, Blackpool
  - Barts Health NHS Trust, London